CLINICAL TRIAL: NCT06060054
Title: Continuous Measurement of Glymphatic Activity in the Human Brain During Sleep-Wake States
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Applied Cognition (Industry)
Collaborators: University of Washington (Other); Oregon Health and Science University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: AC.2022.03
Record Dates: First submitted 2023-09-16; First posted 2023-09-29 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Cross-over randomized study
Who Masked: Outcomes Assessor
Masking Description: Visit type was masked to neuroimaging assessors and blood biomarker analysis laboratory.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Sleep Opportunity (Experimental): Overnight sleep wearing the device
  Interventions: Diagnostic Test: Device measurements
- Sleep Deprivation (Experimental): Overnight awake wearing the device
  Interventions: Diagnostic Test: Device measurements

INTERVENTIONS:
Diagnostic Test: Device measurements — Overnight device measurements

SUMMARY:
This is a cross-over randomized study to validate the Sponsor investigational medical device against measurements of glymphatic function from MRI-based neuroimaging, EEG, blood biomarkers and cognitive tests in healthy older volunteers.

DETAILED DESCRIPTION:
The study population will consist of healthy individuals, ages 50 to 65, that are cognitively normal and do not have a medical history of neurological or sleep disorder, cardiovascular disease, hypertension, or diabetes. The objectives of this study are to define whether sleep- and wake-associated device measurements (i) faithfully reflect glymphatic function measured by non-invasive MRI measures of glymphatic function; (ii) replicate pre-clinical findings between sleep EEG power bands and glymphatic flow; (iii) predict plasma levels of Alzheimer's disease (AD)-related biomarkers; and (iv) predict morning cognitive performance.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have a Montreal Cognitive Assessment (MoCA) score at least 26.
2. Participants must have a Geriatric Depression Scale (GDS) 15-item score of 4 or less.

Exclusion Criteria:

1. Participants with a formal diagnosis of any sleep disorder (e.g., sleep apnea on positive-airway-pressure (PAP) therapy, insomnia, restless leg syndrome, circadian rhythm sleep disorder, parasomnia).
2. Participants with a history of significant neurological disease or history of epilepsy.
3. Participants with cardiovascular disease or cardiovascular risk factors (smoking or hypertension).
4. Participants with diabetes.
5. Participants with traumatic brain injury, or serious mental illness including bipolar disorder, schizophrenia, major depressive disorder or post-traumatic stress disorder.
6. Participants who have taken in the past 30 days prescribed or over-the-counter (OTC) stimulants, sleeping medications, or psychiatric medications including antidepressants.
7. Participants who consume more than 400 mg/day of caffeine. Participants will be required to not consume caffeine beginning 12pm on the day-of the sleep study.
8. Female Participants who consume more than 3 alcoholic drinks on any day or more than 7 drinks per week. Male participants who consume more than 4 alcoholic drinks on any day or more than 14 drinks per week.
9. Participants who have or will have travelled across time zones 10 days prior to either Study Visit or whose first and second Study Visits span Daylight Savings time change (November 6, 2022).
10. Participants with travel plans or conflicts that would prevent them from either Study Visit.
11. Participants who are enrolled in other research studies and are receiving an investigational drug within 30 days of the planned start date.
12. Participants who have any condition that, in the opinion of the Sponsor Principal Investigator, would compromise the well-being of the participant or the study or prevent the participant from meeting or performing study requirements.
13. Participants with absolute or relative contraindications to MRI imaging based on current up-to-date screening questionnaires including claustrophobia, inability to lie still on their back for 30-45 minutes or require sedation prior to the MRI.
14. Participants with a head circumference greater than 60 cm that would prevent use of a high-resolution 64 channel MRI head coil required for this study
15. Participants who have a pre-planned surgery or medical procedure that would interfere with the conduct of the study.
16. Participants who have an implanted medical device or contraindications that would exclude MRIs
17. Participants with a serious infection requiring medical attention in the past 30 days

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-05-10 (Actual); Study Completion 2023-05-10 (Actual)

PRIMARY OUTCOMES:
MRI | Immediately before and immediately after the intervention
  Define whether sleep- and wake-associated device measurements (impedances in milli-ohms) faithfully reflect glymphatic function measured by non-invasive MRI measures of glymphatic function: (i) diffusion-based intravoxel incoherent motion (IVIM)-MRI (long-distance water transport) (diffusion signal, a.u.), (ii) fast functional MRI (f-MRI) low-frequency vasomotor oscillations, Hz, (iii) T1/FLAIR-based assessment of MRI-visible perivascular spaces (MV-PVS) that are structural indicators of perivascular impairment, (a.u.); (iv) multi-echo arterial spin-labeling (ME-ASL)-MRI (glial-vascular water transport) (flow in ml/sec); (v) and phase-contrast (PC)-MRI (aqueductal cerebral spinal fluid (CSF) flow) (flow in ml/sec).

SECONDARY OUTCOMES:
Sleep EEG | During the intervention
  Correlations between device overnight measurements (impedances in milli-ohms) and overnight recorded EEG power bands (relative delta, theta, alpha and beta power in %) replicate pre-clinical correlations of glymphatic flow (measured using 2-photon microscopy in a.u.) and EEG power bands (relative delta, theta, alpha and beta power in %).
Blood biomarkers | Immediately before and immediately after the intervention
  Device overnight measurements predict overnight changes in amyloid beta40, beta42, n-tau 181, n-tau 217, p-tau 181, p-tau 217 blood biomarkers.
Cognitive function | Immediately after the intervention
  Device overnight measurements predict morning cognitive performance based on aggregated standardized scores (mean of 0 and standard deviation of 1) of Trail Making Tests A&B (time in seconds), symbol digit modality test (SDMT) (number correct), psychomotor vigilance test (PVT) (mean and standard deviation of reaction time) and digits forward recall (maximum number of correctly recalled digits).

CONTACTS AND LOCATIONS:
Overall Officials: Paul Dagum, MD PhD, Principal Investigator — Applied Cognition, Inc.
Locations (1):
- University of Washington Department of Radiology (DISC), Seattle, Washington, United States